CLINICAL TRIAL: NCT02812147
Title: Effect of L-Dihydoxyphenylserine (L-DOPS, Northera) a Central and Peripheral Norepinephrine Agent on Locomotion, Postural Stability (Balance), and Fall Risk Reduction in Parkinson Disease (PD)
Brief Title: Effect of L-Dihydoxyphenylserine on Locomotion, Postural Stability, and Fall Risk Reduction in Parkinson Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Pam Dewey, Research Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PHX15BN108
Record Dates: First submitted 2016-05-25; First posted 2016-06-24 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Parkinson Disease
Keywords: L-dihydoxyphenylserine; L-DOPS; Northera
MeSH Terms: conditions — Parkinson Disease | interventions — Droxidopa; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-DOPS (Active Comparator): All participants will be on levodopa/carbidopa, and may be on additional dopaminergic drugs including dopamine agonists and/or monoamine type B oxidase inhibitors or amantadine. L-dihydoxyphenylserine will be added, administered as an oral capsule 3 times a day for 4 months. Dosing will begin at 100 mg of L-DOPS three times per day and titrated upward, by 100 mg three times a day, as tolerated. Tolerability will be evaluated based upon questionnaires, patient interviews, vital signs and investigator examination. In order to participate in the study, all subjects must be able to tolerate a minimum tolerated dose of 400 mg three times per day (1200mg/day). Subject maximum dose will be 600 mg three times per day (1800mg/day). Patients will be maintained on this dose for 4 months (until the cross-over). After a 7-day washout, participants will cross over to the Placebo arm.
  Interventions: Drug: L-DOPS
- Placebo (Placebo Comparator): All participants will be on levodopa/carbidopa, and may be on additional dopaminergic drugs including dopamine agonists and/or monoamine type B oxidase inhibitors or amantadine. Placebo will be added, administered as an oral capsule 3 times a day for 4 months. Dosing will begin at 100 mg of placebo three times per day and titrated upward, by 100 mg three times a day, as tolerated. Tolerability will be evaluated based upon questionnaires, patient interviews, vital signs and investigator examination. In order to participate in the study, all subjects must be able to tolerate a minimum tolerated dose of 400 mg three times per day (1200mg/day). Subject maximum dose will be 600 mg three times per day (1800mg/day). Patients will be maintained on this dose for 4 months (until the cross-over) After a 7-day washout, participants will cross over to the L-DOPS arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-DOPS — Added as described in the Arm/Group Descriptions.
  Other Names: L-dihydoxyphenylserine; Northera
  Arms: L-DOPS
Drug: Placebo — Added as described in the Arm/Group Descriptions.dded as described in the Arm/Group Descriptions.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
This research study is being done to determine whether treatment with L- Dihydroxyphenylserine (L-DOPS) versus placebo (an inactive substance that looks like study drug) in addition to other Parkinson Disease (PD) drugs will improve balance, walking, and reduce risk of falls and/or severity of falls in PD subjects. The study is also being done to determine the effectiveness, safety, and tolerability of L-DOPS, and whether it will decrease Freezing of Gait (FOG), improve apathy (generalized disinterest) or show a relationship between apathy and slowed movement and fall risk.

DETAILED DESCRIPTION:
Among the top three priorities presented to the National Institute of Neurological Disorders and Stroke (NINDS) Council 22 as final recommendations of critical needs for advancing Parkinson Disease (PD) research in 2014 is to develop effective treatments for dopa-resistant features of PD. These features include symptoms such as gait and balance problems, and freezing of gait leading to falls. In order for these goals to be realized, dysfunctional motor patterns in patients with gait and balance problems need to be accurately defined and assessed using body-fixed sensors and other newer computation technology to enhance sensitivity and specificity of measurement to facilitate long-term follow-up. The proposed research will meet the challenge of determining appropriate intervention (L-DOPS) for dopa-resistant features of PD in improving gait and posture using innovative quantitative analyses derived from body-worn sensors. Injuries associated with fall incidences continue to pose a significant burden to persons with Parkinson's disease (PD) both in terms of human suffering and economic losses. Annual fall incidence rates range from 50-70% of patients with PD. Recurrent falls especially, are a major cause of disability in PD. The resulting loss of independence and treatment costs add substantially to the healthcare expenditures in PD which was estimated to be $27 billion annually2. This number may rise substantially in the coming decades as the entire US population ages. Any intervention that is cost effective at reducing fall risk could have important benefits for patients and families, and for the entire healthcare system. In this study, we will determine whether treatment with L- Dihydroxyphenylserine (L-DOPS, Northera) in addition to dopaminergic drugs will improve postural stability and activity of daily living, and reduce fall risk and/or severity of falls in PD patients.Falls, early in PD (within 5 years of diagnosis) probably arise from slowed locomotion. Slowed locomotion is corrected by dopaminergic drugs, hence falls early in PD are decreased by such drugs. Later in PD (5 or years after diagnosis) falls, recurrent falls, occur despite such drugs. There is evidence that falls late in PD occur because of impaired postural stability which does not respond to dopaminergic drugs or may be made worse by such drugs. A single fall, although serious, may be only partly related or even unrelated to PD. "Serious fall" is defined as: all four limbs hit the ground, the skull hits the ground, or there is soft tissue or bone injury. However, some people with PD fall repeatedly. In such patients the role of impaired postural stability was stressed. Although the mechanisms underlying impaired postural stability are not well-known in patients with PD, attention is focused on the noradrenergic system. L-DOPS, a drug that enhances norepinephrine levels in the peripheral and central nervous systems, has been shown to moderate orthostatic hypotension, and often improve some PD symptoms. There is evidence that mechanisms related to norepinephrine centers in the basal forebrain and the locus ceruleus play a role in maintaining postural stability in activities of daily living. They may play a role in preventing or ameliorating falls and freezing of gait. FOG is a major problem in patients with PD who fall. There is evidence that L-DOPS, by improving FOG, decreases risk of falls. Additionally, evidence indicates that L-DOPS decreases falls independent of improving FOG. Apathy, a major and disabling non-motor symptom of PD, may be related to decreased central norepinephrine levels. Apathy may be associated with slowed movements and slowed movements may contribute to falls. There is evidence that L-DOPS, by increasing central norepinephrine, may improve apathy and this may result in a decreased risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Subject has voluntarily signed and dated an informed consent form (ICF) prior to any participation in the study.
* Hoehn and Yahr Stage II, III, IV in an "on" state.
* Fell more than twice in past year.
* Montreal Cognitive Assessment (MOCA) score ≥ 24.
* Stable dose of levodopa, dopamine agonist, amantadine, and/or monoamine oxidase B inhibitor, i.e. unchanged for 3 months.
* Subject is ambulatory and able to walk ≥ 10 meters with/without the use of an assistive device.

Exclusion Criteria:

* Patients with atypical Parkinson disorders that result in a high number of falls.These disorders include: Progressive Supranuclear Palsy (PSP), Multiple System Atrophy (MSA), Primary Freezing of Gait (PFG), and Corticobasal Degeneration.
* Patients with dementia MOCA ≤ 23.
* Patients with symptomatic Orthostatic Hypotension being treated with midodrine, fludrocortisone or L-DOPS.
* Patients with uncontrolled hypertension.
* Patients with known allergies to L-DOPS or its excipients.
* Patients with major orthopedic problems of their hips or knees, and patients who need hip or knee replacements.
* Patient with schizophrenia, a schizo-affective disorder, or a bipolar disorder.
* Patients with hallucinations, psychoses, or delusions.
* Patients with a history of recent stroke or myocardial infarction.

Ages: 30 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Motor Score | 4 months
  Measured with United Parkinson's Disease Rating Scale (Part III 0-45) in the medication state of "on", "off", or both.
Balance Score | 4 months
  Measured using Barrow Neurologic Institute (BNI) Balance Scale 0-20, in the medication state of "on", "off", or both.
Postural Stability | 4 months
  Measured using a NeuroCom Equitest System, which tests sensory organization, motor control time, and postural sway measures, in the medication state of "on", "off", or both.
Dynamic Stability | 4 months
  Dynamic stability is measured by wearable devices (Inertial Measurement Units) that collect gait parameters during gait and postural transitions,in the medication state of "on", "off", or both.
Falls | 4 months
  Incidence of falls is self-report, in the medication state of "on", "off", or both.

SECONDARY OUTCOMES:
Freezing of Gait (FOG) | 4 months
  Measured using United Parkinson's Disease Rating Scale (FOG subtests 2.13 and 3.11) 0-8, in the medication state of "on", "off", or both.
Apathy | 4 months
  Measured using Apathy in Parkinson's Disease Questionnaire 0-42, in the medication state of "on", "off", or both.
Orthostatic Hypotension | 4 months
  Measured using Orthostatic Hypotension Symptom Assessment 0-10,in the medication state of "on", "off", or both.

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Lieberman, MD, Principal Investigator — Barrow Neurological Institute/St. Joseph's Hospital and Medical Center
Locations (1):
- Barrow Neurological Institute/St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No